CLINICAL TRIAL: NCT06899386
Title: A Randomized Prospective Clinical Study Evaluating the Effectiveness of the BEAUTIBOND XTREME Adhesive System Using Different Bonding Techniques in Class I and II Restorations: One-Year Results.
Brief Title: Evaluation Of the BEAUTIBOND XTREME Adhesive in Class I and II Restorations: One-Year Results.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Larissa Fernanda Pereira, Co-Author, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 61246422.4.0000.5498
Record Dates: First submitted 2025-03-14; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Adhesive System
Keywords: adhesive system; randomized clinical trial

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- CI: Class I cavities restored with the total acid-etching technique. (Experimental): Class I cavities restored with the total acid-etching technique.
  Interventions: Other: Group CI and CII - BeautiBond Xtreme (total-etch technique) + Beautifil LS
- CII: Class II cavities restored with the total acid-etching technique. (Experimental): Class II cavities restored with the total acid-etching technique.
  Interventions: Other: Group CI and CII - BeautiBond Xtreme (total-etch technique) + Beautifil LS
- TI: Class I cavities restored with the self-etching technique. (Experimental): Class I cavities restored with the self-etching technique.
  Interventions: Other: Group TI and TII - BeautiBond Xtreme (self-etch technique) + Beautifil LS:
- TII: Class II cavities restored with the self-etching technique. (Experimental): Class II cavities restored with the self-etching technique.
  Interventions: Other: Group TI and TII - BeautiBond Xtreme (self-etch technique) + Beautifil LS:
- TIII: Class I cavities restored with the select-etching technique. (Experimental): Class I cavities restored with the select-etching technique
  Interventions: Other: Group TIII and TIV - BeautiBond Xtreme (selective acid-etch technique) + Beautifil LS
- TIV: Class II cavities restorCed with the select-etching technique. (Experimental): Class II cavities restorCed with the select-etching technique.
  Interventions: Other: Group TIII and TIV - BeautiBond Xtreme (selective acid-etch technique) + Beautifil LS

INTERVENTIONS:
Other: Group CI and CII - BeautiBond Xtreme (total-etch technique) + Beautifil LS — the enamel was etched for 30 seconds and the dentin for 15 seconds using 35% phosphoric acid gel (Ultradent). The acid was then rinsed off, and excess moisture was removed with an air spray. To protect the dentin during air blasting, an absorbent paper was held over it using clinical tweezers, ensuring a whitish appearance for the enamel and slightly moist dentin. Excess water on the cotton roll was dried as well. The BeautiBond Xtreme adhesive system was applied without any waiting time, followed by a gentle air spray for 3 seconds and then a strong air blast to ensure solvent evaporation. Finally, the adhesive was light-cured for 5 seconds using a LED photopolymerizer (Gran Valo LED Curing Light, Ultradent).
  Other Names: total-etch technique
  Arms: CI: Class I cavities restored with the total acid-etching technique.; CII: Class II cavities restored with the total acid-etching technique.
Other: Group TI and TII - BeautiBond Xtreme (self-etch technique) + Beautifil LS: — no acid etching was performed on either the enamel or dentin. The BeautiBond Xtreme adhesive system was applied immediately, without any waiting time, followed by a gentle air spray for 3 seconds and then a strong air blast to ensure solvent evaporation. The adhesive was then light-cured for 5 seconds using a LED photopolymerizer (Gran Valo LED Curing Light, Ultradent).
  Other Names: self-etch technique
  Arms: TI: Class I cavities restored with the self-etching technique.; TII: Class II cavities restored with the self-etching technique.
Other: Group TIII and TIV - BeautiBond Xtreme (selective acid-etch technique) + Beautifil LS — the enamel was etched for 15 seconds using 35% phosphoric acid gel (Ultradent). The acid was then rinsed off, and excess moisture was removed with an air spray, leaving the enamel with a whitish appearance. Excess water on the cotton roll was also dried. Next, the BeautiBond Xtreme adhesive system was applied immediately, without any waiting time, followed by a gentle air spray for 3 seconds and then a strong air blast to ensure solvent evaporation. The adhesive was then light-cured for 5 seconds using a LED photopolymerizer (Gran Valo LED Curing Light, Ultradent).
  Other Names: selective acid-etch technique
  Arms: TIII: Class I cavities restored with the select-etching technique.; TIV: Class II cavities restorCed with the select-etching technique.

SUMMARY:
This randomized clinical trial aimed to evaluate the performance of the Beautibond Xtreme adhesive system under different bonding techniques. Patients over 18 years old with restorative needs were selected, and 152 teeth were randomized using the "Research Randomizer Program" for allocation into control groups (CI - Class I restoration with total-etch conditioning; CII - Class II restoration with total-etch conditioning) and test groups (TI - Class I restoration in self-etch mode; TII - Class II restoration in self-etch mode; TIII - Class I restoration with selective enamel etching; TIV - Class II restoration with selective enamel etching). The restorations were evaluated (USPHS criteria) regarding anatomy, integrity, marginal staining, color, roughness, secondary caries lesions, postoperative sensitivity, and retention. Two calibrated examiners (Kappa test 0.84), blinded to the treatments, conducted evaluations for up to one year.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Occlusal stability supported by molars, Presence of at least one premolar or one molar with Class I/II cavities suitable for direct restoration or restoration replacement
* Ability to attend evaluation and regular maintenance appointments
* No clinical symptoms or radiographic signs suggesting pulp involvement
* No periodontal pockets or compromised biological space invasion
* Ability to perform absolute isolation of the operative field and subsequent restoration of the cavity with composite resin
* Active carious lesion
* Occlusal/occlusoproximal surface of molars and premolars, with a radiographic image showing shallow, medium, or deep dentin involvement, which is preventing the patient from effectively controlling bacterial biofilm, or showing some type of sensitivity
* Cavity preparation margins (cavosurface) in enamel or dentin.

Exclusion Criteria:

* Poor oral hygiene control
* Patients undergoing orthodontic treatment
* Pregnant or lactating women
* Oral complications such as: bruxism, other parafunctional habits reinforcing the diagnosis of TMD (temporomandibular disorders), periodontal problems
* Pregnant or breastfeeding women
* Presence of uncontrolled systemic diseases
* Patients at high risk for caries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Anatomic Form | baseline, six months, and one year.
  The anatomic form of the restoration was evaluated according to the modified United States Public Health Service (USPHS) criteria at baseline, six months, and one year. Restorations were classified as Alpha (continuity of the restoration with the existing anatomic form), Bravo (continuity of the restoration with partial degradation but clinically acceptable), or Charlie (continuity of the restoration compromised, requiring replacement).
Marginal Adaptation | baseline, six months, and one year.
  Marginal adaptation was visually analyzed using an explorer to detect crevices or marginal failures. Classifications included Alpha (no visible evidence of a crevice along the margin), Bravo (visible evidence of a crevice along the margin where the explorer can penetrate or catch), and Charlie (the explorer penetrates the crevice, exposing dentin or base).
Marginal Discoloration | baseline, six months, and one year.
  Marginal discoloration was assessed by recording any color changes at the interface between the restoration and tooth structure. Restorations were classified as Alpha (no visible discoloration), Bravo (discoloration present but not penetrating along the margin in a pulpal direction), or Charlie (deep discoloration penetrating along the margin toward the pulp).
Secondary Caries | baseline, six months, and one year.
  The presence of secondary caries was clinically and radiographically evaluated throughout the study. Restorations were classified as Alpha (no evidence of secondary caries) or Charlie (evidence of secondary caries around the restoration, requiring replacement).
Color Match | baseline, six months, and one year.
  Color match was evaluated by comparing the restoration to the adjacent tooth structure in terms of color and translucency. Classifications included Alpha (color and translucency compatible with the tooth structure), Bravo (color and translucency mismatch within the acceptable range), and Charlie (color and translucency mismatch outside the acceptable range).
Postoperative Sensitivity | baseline, six months, and one year.
  Postoperative sensitivity was assessed through patient reports at different study periods. Classifications included Alpha (no postoperative sensitivity after the restorative procedure and throughout the study), Bravo (slight sensitivity at any stage of the study), and Charlie (severe sensitivity at any stage of the study).
Surface Texture | baseline, six months, and one year.
  The surface texture of the restoration was visually and tactilely evaluated using an explorer. Restorations were classified as Alpha (no surface defects), Bravo (minimal surface defects), or Charlie (severe surface defects on the restoration).
Retention | baseline, six months, and one year.
  Retention was evaluated by verifying the presence of the restoration over time. Classifications included Alpha (no loss of restorative material) and Charlie (fracture and/or total loss of the restorative material).

CONTACTS AND LOCATIONS:
Locations (1):
- Ribeirão Preto School of Dentistry of the University of São Paulo (FORP-USP), Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes